CLINICAL TRIAL: NCT04388865
Title: Clinical Hovering to Improve Patient Engagement in Inflammatory Bowel Disease
Brief Title: Patient Automated Text Hovering for IBD
Acronym: PATH-IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shivan J Mehta, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 842733
Record Dates: First submitted 2020-05-07; First posted 2020-05-14 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Behavioral Economics; Patient Engagement; Remote Monitoring
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Patient Participation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Usual Care
  Interventions: Behavioral: Control
- Clinical Hovering (Experimental): Remote monitoring with feedback to social support
  Interventions: Behavioral: Text-based Clinical Hovering

INTERVENTIONS:
Behavioral: Control — Subjects will engage with their providers as is standard of care.
  Arms: Control
Behavioral: Text-based Clinical Hovering — Subjects will receive remote monitoring via text messaging of clinical symptoms and medication adherence reminders with feedback to social support.
  Arms: Clinical Hovering

SUMMARY:
This is a 2-arm randomized trial aimed at leveraging behavioral science principles to improve patient engagement between office visits among patients with inflammatory bowel disease (IBD).

DETAILED DESCRIPTION:
Crohn's Disease (CD) and Ulcerative Colitis (UC), collectively known as inflammatory bowel disease (IBD), are common chronic gastrointestinal diseases with significant morbidity and decreased quality of life. Care for patients with IBD has been transformed by biologic therapies which dramatically improve inflammation and clinical outcomes. As they are delivered through infusion or injection with long intervals between doses, it can be challenging for patients to maintain adherence due to systems issues such as prior authorization and site of service limitations, in addition to traditional reasons for non-adherence such as inertia and present-time bias. Despite evidence that high adherence is needed for effectiveness, estimates are as low as 66%.

Preliminary observations and interviews show that an important gap for providers is lack of knowledge of how their patients are doing between visits. Specifically, patients may not adhere to necessary therapy, and physicians are unaware of changes in course of the disease. A large cross-sectional study has shown that patient-reported outcomes are associated with control of the disease, but serially monitoring these measures has not been tested prospectively. A prior study found that assessing symptoms weekly is highly correlated with information collected with a more cumbersome daily diary. This may provide additional data to clinicians to better manage symptoms and therapy.

Text messaging is an attractive tool to engage with patients due to the high prevalence of cell phones. The investigators will develop and test a new IBD hovering program that improves the care of patients between office visits. The investigators will enroll patients prescribed biologic therapy and provide text message reminders about scheduled infusions or injections that incorporate behavioral science principles such as anticipated regret, precommitment, and reciprocity. The investigators will also have the patient identify a friend or family member to serve as a support partner to encourage adherence and provide assistance as needed. The platform will communicate with patients weekly to ask about the course of their symptoms, send messaging to the feedback partner, and send alerts to physicians as needed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's Disease or Ulcerative Colitis
* Has had at least 2 visits with Penn Gastroenterology in the past 2 years
* Currently prescribed a biologic therapy (infliximab, adalimumab, ustekinumab, certolizumab, golimumab, or vedolizumab). Of note, this study is not limited to new initiators of these medications.

Exclusion Criteria:

* Patients will be excluded if they do not have a phone with text messaging.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) response | 4 months
  The change in patient response to the Short Inflammatory Bowel Disease Questionnaire (SIBDQ), which is a 10 question validated instrument to measure quality of life in IBD patients.

SECONDARY OUTCOMES:
Patient Satisfaction | 4 months
  Patient satisfaction, adapted from the CACHE questionnaire, will be measured by the percent who agree/totally agree (scored as 1 or 2 on a scale of 1-5) to each survey question. A net promoter score (scored as percent 9 or 10 minus percent 1-6 on a scale of 1-10) will also be calculated for the intervention group only.
Medication Adherence | 4 months
  Medication adherence will be measured as show rate for infusions and percent dispensed by pharmacy for injectables based on chart review at pre- and post-intervention, along with the change in percent reported adherence at the baseline and post-study survey.

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No